CLINICAL TRIAL: NCT06928272
Title: LC-REVITALIZE - A Long Covid Repurposed Drug Study
Brief Title: Long Covid (LC)-REVITALIZE - A Long Covid Repurposed Drug Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Douglas D. Fraser (Other)
Responsible Party: Sponsor-Investigator, Douglas D. Fraser, MD, PhD, FRCPC, Professor and Clinician Scientist, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LC-Revitalize
Record Dates: First submitted 2025-04-03; First posted 2025-04-15 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Long COVID
Keywords: Post-Covid-19 Condition; Covid-19; SARS-CoV-2
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — pirfenidone; upadacitinib

STUDY DESIGN:
Intervention Model Description: This study employs an adaptive, platform study design, allowing for flexibility in the evaluation and management of various interventions within an overarching core protocol to identify the best performing drug. The adaptive framework is designed to maximize efficiency, improve participant outcomes, and accelerate decision-making based on pre-specified criteria.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pirfenidone (Experimental): 267mg pirfenidone tablets, over encapsulated in hard-gelatin capsules
  Interventions: Drug: Pirfenidone
- Placebo for Pirfenidone (Placebo Comparator): Hard-gelatin capsules that are made to look and feel like the pirfenidone over encapsulated drug
  Interventions: Drug: Placebo for pirfenidone
- Upadacitinib (Experimental): 15 mg upadacitinib tablets, over encapsulated in hard-gelatin capsules
  Interventions: Drug: Upadacitinib
- Placebo for Upadacitinib (Placebo Comparator): Hard-gelatin capsules that are made to look and feel like the upadacitinib over encapsulated drug
  Interventions: Drug: Placebo for upadacitinib

INTERVENTIONS:
Drug: Pirfenidone — Initial dose titration:
  First week (days 1-7): 1 capsule (267 mg), 3 times daily (801 mg/day)
  Second week (days 8-14): 2 capsules (534 mg), 3 times daily (1602 mg/day)
  Maintenance dose:
  Third week and thereafter (days 15-90): 3 capsules (801 mg), 3 times daily (2403 mg/day)
  Other Names: Esbrit
  Arms: Pirfenidone
Drug: Placebo for pirfenidone — First week (days 1-7): 1 capsule, 3 times daily
  Second week (days 8-14): 2 capsules, 3 times daily
  Third week and thereafter (days 15-90): 3 capsules, 3 times daily
  Arms: Placebo for Pirfenidone
Drug: Upadacitinib — 1 capsule (15 mg), once daily for 90 days
  Other Names: Rinvoq
  Arms: Upadacitinib
Drug: Placebo for upadacitinib — 1 capsule, once daily for 90 days
  Arms: Placebo for Upadacitinib

SUMMARY:
The Long-Covid (LC)-Revitalize clinical study is testing repurposed drug treatments for Long Covid, involving adult participants from Brazil, Canada, Italy, Uganda, the United States, and Zambia. To qualify, participants must have had Covid-19 and experienced Long Covid symptoms for at least three months. The main goal of the study is to determine whether the drug treatments can improve symptoms in five key areas: 1) fatigue, 2) breathing, 3) memory, thinking, and communication, 4) muscle and joint pain, and 5) circulation. A secondary goal is to assess changes in the body, such as reducing inflammation, as well as to confirm the safety and tolerability of the treatments. In the first phase, 348 participants will take either one of two existing medications (upadacitinib or pirfenidone) or a placebo (a pill with no active ingredient) for three months. Although these medications are not yet approved for Long Covid, they are authorized for use in treating other health conditions. This study is adaptive, meaning it may adjust based on early results. In the second phase, the study could continue testing the most effective drug(s) against a placebo with new participants, explore combinations of drugs to see if they improve results, or discontinue the drugs if they prove ineffective or unsafe and test alternative treatments.

DETAILED DESCRIPTION:
Long Covid represents a significant public health challenge, yet effective treatments remain elusive due to the disease's heterogeneity, limited clinical data, and inconsistent methodologies. A previous analysis of clinical and proteomic data from 1,028 subjects diagnosed with Long Covid across three continents (The LC-Optimize Study) suggests that certain repurposed medications may offer potential therapeutic benefits.

Drug repurposing is based on the principle that many drugs interact with multiple molecular targets and mechanisms of action, potentially extending their effects beyond their original intended use. This phenomenon arises from the complex nature of biological systems and the interactions between drugs and various cellular components, which our research pipeline is designed to identify.

A key advantage of repurposed drugs is that they already have established safety and toxicity profiles, are approved by regulatory authorities, and can therefore expedite clinical trials with sufficient supporting data and justification.

This is a Phase III, double-blind, placebo-controlled, multi-arm platform study that will enroll participants from Brazil, Canada, Italy, Uganda, Zambia, and the United States. The first phase of the study will enroll approximately 348 participants globally, all of whom must have previously tested positive for SARS-CoV-2 and have been experiencing Long Covid symptoms for three months or more. A second phase will follow, guided by the results of the first phase and determined through an interim analysis. This phase, which will occur after a protocol amendment, may involve continued testing of one or both repurposed drugs, combination treatments with an additional repurposed drug, or the introduction of a completely new repurposed drug.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must meet all the following inclusion criteria:

1. Adults ≥ 18 years of age and ≤ 65 years of age
2. Previous Covid-19 (SARS-CoV-2 infection) within the past four years, as determined by the site investigator using the following certainty scale (based on available clinical history and/or serologic data):

3 - Confirmed Infection (PCR or n-Capsid Test): Prior positive nasopharyngeal or salivary PCR test for Covid-19 (documented proof and/or verbal confirmation by participant) or has positive nucleocapsid antibodies results.

2 - Probable Infection (Antigen Test): Participant verbally confirms a prior positive rapid antigen test without PCR confirmation.

1 - Possible Infection (Viral Syndrome and Epidemiological Link): Participant verbally confirms experiencing symptoms consistent with Covid-19 infection and has an epidemiological link (i.e., exposure to a confirmed case) without any positive testing.

3. Persistent or new symptoms diagnosed as "Long Covid" as defined by the World Health Organization; "the continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection (Covid-19), with these symptoms lasting for at least 2 months with no other explanation". This diagnosis may come from a healthcare professional experienced in Long Covid diagnosis, or the site investigator. These symptoms must be present for more days than not and must not have been present prior to the onset of SARS-CoV-2 (Covid-19) infection.

4. At the time of screening, participants should be experiencing at least one of the following self-reported symptoms or symptom clusters. Participant has self-reported issues with:

1. Fatigue
2. Breathing
3. Circulation
4. Memory, thinking, and/or communication
5. Muscles and/or joints

   These five symptoms or symptom clusters were selected based on unpublished data from the National Institutes for Health and Care Research (NIHR, United Kingdom) and their alignment with five validated SBQ scales. The selection was driven by their prevalence and their significant impact on quality of life as reported in symptom assessments.

   5. Participant has the ability and is willing to follow study procedures throughout the study

   6. Participant can provide informed consent

   Exclusion Criteria:

   Participants who have any one or more of the following criteria at the time of enrollment will be excluded:
   1. Participants who do not meet the criteria outlined above
   2. Participants who are unable to provide their informed consent
   3. Participants who are pregnant, lactating, or plan to become pregnant during the time of the study
   4. Persons of childbearing potential who are unwilling or unable to abstain from sex or to use at least one acceptable method of contraception from the time of screening through at least 30 days after the end of the study intervention period. Acceptable methods include barrier contraceptives (e.g., condoms or diaphragm) with spermicide, intrauterine devices (IUDs), hormonal contraceptives, oral contraceptive pills, and surgical sterilization. Participants unwilling to be counseled about the risks related to pregnancy or breastfeeding will also be excluded.
   5. Male participants must take precautions to avoid impregnating a female while participating in this study. If a male participant's partner can become pregnant, she must use an effective and reliable form of birth control, as listed above, during the study and for 30 days after the male participant's last dose of the investigational product. Additionally, male participants must agree to use a latex condom during sexual activity with partners who could become pregnant.
   6. eGFR <30 mL/min/1.73m2
   7. Moderate to severe liver dysfunction, defined as Bilirubin > 1.5 x ULN or AST or ALT > 2 x ULN
   8. Hemoglobin (Hbg) < 8.0 g/dL
   9. Absolute neutrophil count (ANC) below 1,000 cells/mm³, confirmed with repeat testing
   10. Absolute lymphocyte count (ALC) below 500 cells/mm³
   11. Alkaline phosphatase (ALP) levels equal to or greater than three times the upper limit of normal (ULN)
   12. Creatine phosphokinase (CPK) levels equal to or greater than three times the ULN
   13. Platelet count below 100,000 cells/mm³, confirmed with repeat testing
   14. Platelet count above 500,000 cells/mm³, confirmed with repeat testing
   15. Total fasting cholesterol levels of 280 mg/dL or higher, confirmed with repeat testing
   16. Fasting low-density lipoprotein (LDL) levels of 180 mg/dL or higher, confirmed with repeat testing
   17. A personal or family history of long QT syndrome or an electrocardiogram (ECG) during screening showing a corrected QT interval (QTc) of 500 milliseconds or greater, calculated using Fridericia's formula
   18. Participants with HIV diagnosis
   19. Participants with active hepatitis B or C diagnosis. Note: treated or cleared hepatitis C is not exclusionary.
   20. Active herpes zoster infection (visible skin lesions) within 3 months prior to screening, or any history of disseminated or complicated herpes zoster or herpes simplex infection (e.g., VZV encephalitis)
   21. Participants with active or latent tuberculosis
   22. Immunocompromised status, as determined by the investigator, that places the participant at an unacceptable risk for study participation
   23. Active malignancy or lymphoproliferative disorder that has not been in remission for at least five years. Localized non-melanoma skin cancers that have been definitively treated are not exclusionary.
   24. Positive SARS-CoV-2 test in the last 30 days or symptomatic with Covid-19 like illness
   25. Previous admission to an intensive care unit (ICU) for the treatment of acute COVID-19 infection
   26. Any history of deep venous thrombosis, pulmonary embolism, unstable angina, atrial fibrillation, ventricular fibrillation, or myocardial infarction or stroke
   27. History of sepsis or a significant viral, bacterial, fungal, or parasitic infection within 30 days prior to enrollment, as determined by the investigator.
   28. Use of one or more of the study drugs within 30 days prior to enrollment for the original indication or other purposes
   29. Known allergic reactions to the components of the study drugs
   30. Any prior exposure to JAK inhibitors
   31. Taking any of the listed medications on the prohibited medications list in Appendix A
   32. Intake or planned consumption of any of the following: Taurine, Curcumin, CoQ10, Creatine, Resveratrol, Fisetin, Nicotinamide mononucleotide (NMN), Nicotinamide adenine dinucleotide (NAD+), Quercetin, Glycine, Spermidine, Arginine alpha-ketoglutarate, Ergothioneine, Alpha Lipoic Acid, Carnitine, Benfotiamine, Carnosine, Crocin, N-acetylcysteine
   33. Covid vaccinations are prohibited within 30 days prior to enrollment
   34. Live vaccine within the 30 days before enrollment or plan to receive live vaccines during the study period
   35. Other vaccines, including influenza vaccine, are prohibited within 14 days of enrollment
   36. Major surgery within 30 days prior to enrollment or plans for major surgery during the study
   37. Any other co-existing medical condition or concomitant medication/therapy that might in the judgment of the study investigators, potentially impact the participant's safety or ability to adhere to the study protocol or interfere with the meaning of the clinical and research measurements as judged by the study investigators
   38. Participation in any clinical study within the last 30 days prior to enrollment
   39. Participants who participated in Phase One of this study (LC-Revitalize) are not eligible to participate in Phase Two
   40. Currently hospitalized and/or incarcerated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Symptom Burden Questionnaire (SBQ) Subscales | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  The aim of this study is to evaluate the efficacy of two repurposed drugs in reducing symptom severity in participants with Long Covid. The change in symptom score (transformed scale of 0-100) from baseline to both the interim and final analyses will be compared across one of the five validated subscales, relative to the placebo.
  This study will utilize five validated subscales: 1) Fatigue, 2) Breathing, 3) Memory, Thinking, and Communication, 4) Muscles and Joints, and 5) Circulation. Each subscale is based on a 4-point ordinal scale that assesses frequency, severity, or interference, or it uses a dichotomous yes/no response. The subscale with the highest symptom burden, determined by the highest transformed symptom score (ranging from 0 to 100, with a higher score indicating greater symptom burden) at baseline, will be selected for evaluating treatment effects.

SECONDARY OUTCOMES:
General participant reported overall well-being using the Patient Reported Outcome Measurement Information System (PROMIS)-29 questionnaire | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  To compare symptom burden of participants with Long Covid treated with study drug versus placebo by measuring the change in total scores of the Patient Reported Outcome Measurement Information System (PROMIS)-29 questionnaire.
  The PROMIS-29 questionnaire consists of 29 items covering an overview of the participant's physical, mental, and social health. Each item is scored on a scale of 1 to 5, with the interpretation of lower scores varying by domain-indicating either better or worse symptom experience.
General participant reported overall well-being using the Generalized Anxiety Disorder (GAD)-7 questionnaire | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  To compare symptom burden of participants with Long Covid treated with study drug versus placebo by measuring the change in total scores of the Generalized Anxiety Disorder (GAD)-7 questionnaire from baseline to the interim and final analyses.
  The GAD-7 questionnaire consists of 7 items relating to the symptoms of stress and anxiety levels. Each item is scored on a scale of 0-3 with higher scores indicating more severe symptoms. Overall scores can range from 0-21 with scores of 5, 10, and 15 taken as the cut-off points for mild, moderate, and severe anxiety, respectively.
General participant reported overall well-being using the Patient Health Questionnaire (PHQ)-9 | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  To compare symptom burden of participants with Long Covid treated with study drug versus placebo by measuring the change in total scores of the Patient Health Questionnaire (PHQ)-9 from baseline to the interim and final analyses.
  The PHQ-9 questionnaire consists of 9 items related to the symptoms of depression. Each item is scored on a scale of 0-3 with higher scores indicating more severe symptoms. Overall scores can range from 0-27 with scores of 5, 10, 15, and 20 taken as cut off points for mild, moderate, moderately severe, and severe depression, respectively.
General participant reported severity of post-exertional malaise (PEM) using the FUNCAP27 questionnaire | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  To compare symptom burden of participants with Long Covid treated with study drug versus placebo by measuring the change in scores of the Functional Capacity (FUNCAP)27 questionnaire from baseline to the interim and final analyses. The FUNCAP27 questionnaire consists of 27 items related to assessing functional capacity and the consequences of performing activities. Each item is scored on a scale of 0-6, with 0 indicating the participant is unable to complete the activity and 6 indicating the activity is unproblematic and does not affect other activities.
Worsening Long Covid Symptoms Measured by SBQ Subscales | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  To assess whether symptom burden worsens in participants with Long Covid treated with study drugs versus placebo, specifically when symptoms are reported across multiple scales indicated by the total number of participants with increased SBQ subscale scores.
  The following SBQ subscales will be used during this study: 1) Fatigue, 2) Breathing, 3) Memory, thinking, and communication, 4) Muscles and joints, and 5) Circulation.
  Each subscale is based on a 4-point ordinal scale that assesses frequency, severity, or interference, or it uses a dichotomous yes/no response. The subscale with the highest symptom burden, determined by the highest transformed symptom score (ranging from 0 to 100, with a higher score indicating greater symptom burden) at baseline, will be selected for evaluating treatment effects.
Quantitative measurement of biomarkers specific to relevant inflammatory pathways and to Long Covid identified previously (The LC-Optimize Study) | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  To measure specific pathophysiological biomarkers of study drugs versus placebo indicated by the normalization of blood biomarkers after treatment in picograms per milliliter (pg/mL).
Exercise capacity assessed by the 6-minute walk test (6MWT) | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  To assess changes in exercise capacity over time of participants with Long Covid treated with study drugs versus placebo. The score is determined by the distance a participant walks in six minutes around the perimeter of a designated circuit.
Safety and tolerability of the study drugs in participants with Long Covid | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  The frequency and severity of adverse events and laboratory abnormalities will be monitored to assess safety and tolerability. A lower incidence and severity will indicate that the drugs are safer and more tolerable.

OTHER OUTCOMES:
A comprehensive OMICS evaluation will be completed to further understand mechanisms of the repurposed drugs | The Phase 1 time frame is from enrollment on Day 1 through to the end of follow-up at Month 6, and the Phase 2 time frame will be determined based on the results of Phase 1.
  Plasma proteomics will be analyzed to assess protein differential expression and signaling pathway mechanisms related to the study drugs. Analyses will focus on the expression normalization of proteins/pathways associated with Long Covid.
  Plasma metabolomics will be analyzed to evaluate metabolic changes and the overall effects of the study drugs. Analyses will focus on the concentration normalization of metabolites linked to the pathophysiology of Long Covid.
  White blood cell (WBC) RNA sequencing will be performed to identify changes in gene expression, offering insight into the body's response to the study drugs. Analyses will focus on transcriptional shifts from baseline to the end of the study.
  Exome sequencing and single nucleotide polymorphism (SNP) analysis will be performed to identify genetic variants that may influence the metabolism and efficacy of the study drugs. This will help identify genetic markers associated with drug non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas D Fraser, MD, PhD, FRCPC, Principal Investigator — Western University
Locations (8):
- Laura Rodriguez Research Institute, San Diego, California, United States
- Ini-Fiocruz, Rio de Janeiro, Rio de Janerio, Brazil
- Canada (2):
  - Institut de Recherches Cliniques de Montréal (IRCM), Montreal, Quebec
  - Centre de Recherche du CHUS (CRCHUS), Sherbrooke, Quebec
- Italy (2):
  - INMI Lazzaro Spallanzani IRCCS, Roma, Roma
  - Sapienza Università di Roma, Roma, Roma
- Joint Clinical Research Centre (JCRC), Kampala, Kampala, Uganda
- University Teaching Hospital, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: No